CLINICAL TRIAL: NCT00421564
Title: A Randomized, Double-Blind, Placebo Controlled Study of the Effect of Danggui Buxue Tang on Menopausal Symptoms and Quality of Life in Hong Kong Chinese Women
Brief Title: Study the Effect of Danggui Buxue Tang on Menopausal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICM/CTS/004
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: Menopause
Keywords: Menopausal; Traditional Chinese Medicine

INTERVENTIONS:
Drug: DBT-Danggui Buxue Tang

SUMMARY:
This study is to examine the effect and safety of the study drug,Danggui Buxue Tang, on menopausal symptoms of hot flushes and sweating and to determine whether the patient's quality of life will be improved.

ELIGIBILITY:
Inclusion Criteria:

* Follicle stimulating hormone (FSH), luteinizing hormone (LH), oestradiol in the menopausal range (FSH>18 IU/L, LH>12.6 IU/L, and E2< 361 pmol/l).
* Patients with amenorrhoea for more than 12 months

Exclusion Criteria:

* Patients with a history of using any form of hormonal replacement therapy within 8 weeks
* Patients with a history of using Chinese medicine or other therapies which may affect the outcome within 8 weeks
* Patients who in the judgment of the investigator will be unable to comply with protocol requirements
* Patients with significant** gastrointestinal, renal, hepatic, bronchopulmonary, neurological, cardiovascular, breast or endometrial carcinoma, or allergic diseases
* Patients with uncontrolled hypertension
* Patients with undiagnosed vaginal bleeding
* Patients with a history of significant drug hypersensitivity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-02; Study Completion 2004-12

PRIMARY OUTCOMES:
The Changes in severity and frequency of hot flushes and sweats.

SECONDARY OUTCOMES:
The Changes in score of the Menopause Specific Quality of Life and the values of various markers of risk for cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Haines, FPOGS, Principal Investigator — Department of Obstetrics & Gynaecology, CUHK
Locations (1):
- Department of Obstetrics & Gynaecology, CUHK, Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Background] Hagstad A, Janson PO. The epidemiology of climacteric symptoms. Acta Obstet Gynecol Scand Suppl. 1986;134:59-65. doi: 10.3109/00016348609157052. PMID 3468732
- [Background] Schneider HP, Gallagher JC. Moderation of the daily dose of HRT: benefits for patients. Maturitas. 1999 Nov;33 Suppl 1:S25-9. doi: 10.1016/s0378-5122(99)00060-2. PMID 10661612
- [Background] Au GK. Evaluation of the benefits and risks of hormone replacement therapy. Hong Kong Med J. 2000 Dec;6(4):381-9. PMID 11177160
- [Background] Blumel JE, Castelo-Branco C, Binfa L, Gramegna G, Tacla X, Aracena B, Cumsille MA, Sanjuan A. Quality of life after the menopause: a population study. Maturitas. 2000 Jan 15;34(1):17-23. doi: 10.1016/s0378-5122(99)00081-x. PMID 10687878
- [Background] Hall G, Pripp U, Schenck-Gustafsson K, Landgren BM. Long-term effects of hormone replacement therapy on symptoms of angina pectoris, quality of life and compliance in women with coronary artery disease. Maturitas. 1998 Jan 12;28(3):235-42. doi: 10.1016/s0378-5122(97)00080-7. PMID 9571599
- [Background] Zhu DP. Dong quai. Am J Chin Med. 1987;15(3-4):117-25. doi: 10.1142/S0192415X87000151. PMID 3425569
- [Background] Davis SR, Briganti EM, Chen RQ, Dalais FS, Bailey M, Burger HG. The effects of Chinese medicinal herbs on postmenopausal vasomotor symptoms of Australian women. A randomised controlled trial. Med J Aust. 2001 Jan 15;174(2):68-71. doi: 10.5694/j.1326-5377.2001.tb143156.x. PMID 11245505
- [Background] Fugh-Berman A. Herb-drug interactions. Lancet. 2000 Jan 8;355(9198):134-8. doi: 10.1016/S0140-6736(99)06457-0. PMID 10675182
- [Background] Chung TK, Yip SK, Lam P, Chang AM, Haines CJ. A randomized, double-blind, placebo-controlled, crossover study on the effect of oral oestradiol on acute menopausal symptoms. Maturitas. 1996 Oct;25(2):115-23. doi: 10.1016/0378-5122(96)01050-x. PMID 8905602